CLINICAL TRIAL: NCT04284033
Title: Evaluation of Extended Wear Infusion Set With 670G Hybrid Closed-Loop Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of sponsor and trial design
Sponsor: Stanford University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Bruce Buckingham, Professor Emeritus, Pediatrics - Endocrinology and Diabetes, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 52526
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard then Extended Infusion Set (Experimental): Participants will start with wearing the standard infusion set for up to 7 days, then switch to the Extended Wear infusion set for up to 7 days, then repeat the cycle for a total of 4 weeks
  Interventions: Device: Extended Wear Infusion Set; Device: Standard Infusion Set
- Extended then Standard Infusion Set (Experimental): Participants will start with wearing the Extended Wear infusion set for up to 7 days, then switch to the standard infusion set for up to 7 days, then repeat the cycle for a total of 4 weeks
  Interventions: Device: Extended Wear Infusion Set; Device: Standard Infusion Set

INTERVENTIONS:
Device: Extended Wear Infusion Set — For two of the 4 weeks, the Extended Wear insulin infusion set will be used
Device: Standard Infusion Set — For two of the 4 weeks, the standard insulin infusion set will be used

SUMMARY:
This is a randomized trial to determine if an extended wear infusion set can be worn for up to 7 days with a hybrid closed-loop system in adult with Type 1 Diabetes

DETAILED DESCRIPTION:
This study will compare use of a standard infusion set with an extended wear infusion set. Subjects will be asked to wear both types of sets twice for up to 7 days, alternating wear of set type over 4 weeks. The order of infusion set wear will be randomized with the first set wear. The investigators aim to see whether there is a benefit to using an extended wear infusion set.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for more than one year, using an insulin infusion pump for at least 6 months, and using the 670G pump for at least 3 months
2. Age ≥18 years
3. Using Novolog or Humalog insulin at time of enrollment
4. For females, not currently known to be pregnant
5. An understanding of and willingness to follow the protocol and sign the informed consent
6. Willing to have photographs taken of their infusion sites
7. Willing to download their 670G pump every week to a research Carelink account
8. Willing to submit a brief online questionnaire at the time of any infusion set failure
9. Able to understand spoken or written English
10. Hemoglobin A1c <8.5% at the time of enrollment
11. Willing to perform three or more fingerstick glucose measurements each day
12. Willing to sign a consent for release of medical information at the time of enrollment
13. Willing to change their infusion pump insulin reservoirs at least every 6 days

Exclusion Criteria:

1. Hypoglycemic seizure or loss of consciousness in the past 6 months
2. Severe episode of DKA in the 6 months prior to study enrollment that was unrelated to an infusion set failure
3. A known cardiovascular disease
4. Active proliferative diabetic retinopathy
5. Known tape allergy
6. Current treatment for a seizure disorder
7. Cystic fibrosis
8. Active infection
9. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol
10. Inpatient psychiatric treatment in the past 6 months
11. Presence of a known adrenal disorder
12. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the last 2 months prior to enrollment in the study
13. Abuse of alcohol
14. History of dialysis, renal failure or known eGFR <60 ml/min/1.73m2
15. Has received a blood transfusion or required treatment for anemia in the three months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Number of infusion set failures due to "unexplained hyperglycemia" | 14 days for each type of infusion set, with each type of infusion set worn twice
  Defined as:
  1. Glucose >250 mg/dL with failure of a correction dose to lower the glucose by 50 mg/dL
  2. Ketones ≥0.6 mg/dL with a glucose reading of >250 mg/dL (in the absence of illness)
  3. Evidence of infection at the infusion site (erythema or induration >1cm in diameter)
  4. Pump occlusion alarm

SECONDARY OUTCOMES:
Duration of infusion set wear | 14 days for each type of infusion set, with each type of infusion set worn twice
  The maximum number of days that 75% of the infusion sets are still working, excluding those that kinked on insertion or were accidentally pulled out.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No